CLINICAL TRIAL: NCT02494531
Title: Illiteracy and Vulnerability to Alzheimer's Disease: Evaluation of Amyloid Pathology by PET Imaging
Acronym: AVILL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P120134
Record Dates: First submitted 2015-05-04; First posted 2015-07-10 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; PET; diagnosis; MCI; illiterate
MeSH Terms: conditions — Alzheimer Disease; Disease; Literacy

ARMS (1):
- Positon Emission Tomographic (PET)-scan (Other): 2 PET-scan: Fluorodeoxyglucose-PET and florbetapir F 18-PET
  Interventions: Radiation: Fluorodeoxyglucose-PET; Radiation: florbetapir F 18-PET

INTERVENTIONS:
Radiation: Fluorodeoxyglucose-PET — Fluorodeoxyglucose-PET performed within 2 months
Radiation: florbetapir F 18-PET — florbetapir F 18-PET performed within 2 months

SUMMARY:
The goal of this study is to improve the diagnosis of Alzheimer's disease (AD) at two different stages (MCI and dementia) in illiterate subjects, using FDG- fluorodeoxyglucose - and florbetapir F 18 -PET imaging. This study will compare amyloid load and cerebral metabolism dysfunction in literate versus illiterate MCI and AD patients.

DETAILED DESCRIPTION:
Illiterate, with a higher rate in the elder and in multi-cultural population reaching, then, 20%. Most of these patients are not usually included in research studies.

Thus, AVILL would specifically focus on lower educated and illiterate patients and on use of PET imaging for early diagnosis. This study would take advantage of the collaboration with the recently launched Memento cohort.

RATIONALE:

1. The diagnosis of AD at the early stages of the disease appears to be crucial. MCI is now considered as the 1st clinical stage of the disease, after a long pre-clinical period.
2. Cognitive reserve modulates the relationship between cerebral lesions and their clinical manifestations by limiting the negative impact of cerebral lesion on cognition. Education is a commonly-used proxy of cognitive reserve. Education interacts with AD pathology such that a greater pathological burden is required to show an effect on cognition among subjects with more education. Lower education and illiteracy are thus considered as risk factor of developing AD
3. Diagnosing MCI and AD in lower educated and illiterate patients is a real challenge because of:

   1. -difficulties in cognitive evaluation which mostly relies on educational background and reading abilities,
   2. -poor adaptation of neuropsychological tests,
   3. -lack of clinical and imaging data concerning these patients, who are often excluded from studies, and poor knowledge of the evolution of the disease from the earlier signs (MCI) to dementia.
4. Quantification of amyloid deposit by PET imaging could therefore be useful for the diagnosis of AD in illiterate patients.

GENERAL OBJECTIVES:

* non educated patient amyloid load could differ from educated patient amyloid load at the same stage of cognitive impairment
* PET amyloid imaging using florbetapir F 18 could detect non educated patients with AD risk at early stage and could help clinical evaluation which is particularly difficult in this population.
* uptake level of florbetapir F 18 could be different in MCI and AD non educated patients compared to educated patients which are the basis of the objectives.

ELIGIBILITY:
Inclusion Criteria:

1. For all patients enrolled in the study:

   * Aged 18 years and above
   * Visual and auditory acuity adequate for neuropsychological testing
   * Having signed an informed consent
   * Being affiliated to health insurance
2. For MCI patients:

   For this group, the criteria are the same as those of Memento but with specially designed neuropsychological tests for illiterate/low educated patients.
   * Performing worse than one standard deviation to the mean (compared to age and educational norms) in one or more cognitive domains (neuropsychological tests battery exploring memory, language, praxis, vision, executive functions); this deviation is required to be documented by tests performed less than 6 months age
   * Clinical dementia Rating scale < or = 0.5
3. For AD patients

   * Fulfilling DSM IV criteria of AD
   * Clinical Dementia Rating scale > 0.5 Patients are defined as "illiterate" having 5 or less years of schooling, and "literate" when having more than 5 years

Exclusion Criteria:

* Being under guardianship
* Residence in skilling nursing facility
* Pregnant or breast feeding women
* Alzheimer's disease caused by gene mutations
* Brain MRI exclusion criteria (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin, or body) or refusing MRI
* Neurological disease such as: treated epilepsy, treated Parkinson's disease, Huntington disease, brain tumour, subdural haematoma, progressive supranuclear palsy, history of head trauma followed by persistent neurological deficits, history of stroke
* Schizophrenia or other psychiatric history (DSM-IV criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-12-12 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the amount of amyloid deposits using florbetapir-18 Fluor-PET between illiterate and literate MCI patients | Within 2 months after inclusion
  Comparison between the 2 groups (educated and non -educated) of florbetapir-18 Fluor Standardized Uptake Values (SUV) ratios (max and mean of SUVr) in MCI patients

SECONDARY OUTCOMES:
Comparison of the amount of amyloid deposits using florbetapir-18 Fluor-PET between illiterate and literate AD patients, | Within 2 months after inclusion
  Comparison of florbetapir-18 Fluor SUV (Standardized Uptake Values) ratios (max and mean of SUVr) in the different groups as defined above
Comparison of the amyloid deposit location between the 2 groups (literate and illiterate) | Within 2 months after inclusion
  Group comparison of qualitative topography of amyloid burden
correlation between amyloid load and metabolism dysfunction using Fluorodeoxyglucose (FDG)-PET in each groups | Within 2 months after inclusion
  Group comparison of topography of amyloid deposit and FDG metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Belin, Dr, Principal Investigator — ASSISTANCE PUBLIQUE HOPITAUX DE PARIS (hospial Avicenne); AMEL OUSLIMANI, PM, Study Director — Assistance Publique - Hôpitaux de Paris, DRCD
Locations (1):
- Hospital Avicenne-Neurology, Bobigny, France